## **SECTION 1: ADMINISTATIVE INFORMATION**

Statistical analysis plan (SAP)



Effect of prothesis and active (PROACT) exercise program in patients with glenohumeral osteoarthritis

Josefine Beck Larsen<sup>1,2</sup>, Theis Muncholm Thillemann<sup>1,2</sup>, Antti P. Launonen<sup>3</sup>, Aleksi Reito<sup>3,4</sup>, Inger Mechlenburg<sup>1,2</sup> and Erik Parner<sup>5</sup>

## **Affiliations:**

<sup>1</sup>Department of Orthopaedic Surgery, Aarhus University Hospital, Aarhus N, Denmark

<sup>2</sup>Department of Clinical Medicine, Aarhus University, Aarhus N, Denmark

<sup>3</sup>Department of Orthopaedic Surgery, Tampere University Hospital, Tampere, Finland

<sup>4</sup>Faculty of Medicine and Health Technology, Tampere University, Tampere, Finland

<sup>5</sup>Department of Public Health, Section for Biostatistics, Aarhus University, Aarhus, Denmark

Chief investigator: Inger Mechlenburg (IM)

Principle Investigator: Josefine Beck Larsen (JBL)

**Senior Biostatistician and:** Erik Parner (EP)

**Analysis Support and Statistical Analyst:** Aleksi Reito (AR)

**Trial registration:** The trial is registered at <u>www.clincaltrials.gov</u> with the number NCT04845074.

**Protocol version:** This document has been written based on the information contained in the trial protocol published in Acta Orthopaedica (1).

Statistical Analysis Plan (SAP) revision history: No revisions have been made.

# Roles, responsibilities, and signatures:

| Role | Name | Date | Signature |
|---------------------|----------------------|------------|------------------|
| SAP author | Josefine Beck Larsen | 02-07-2024 | fife 3. L |
| Senior statistician | Erik Parner | 08-07-2024 | Exil Fames |
| Statistical analyst | Aleksi Reito | 8-7-2024 | |
| Chief investigator | Inger Mechlenburg | 02-07-2024 | Inger Mechhaburg |

#### **SECTION 2: INTRODUCTION**

## **Background**

Glenohumeral osteoarthritis (OA) is characterized by osseous changes, joint incongruence, and capsular thickening (2, 3). Anatomical total shoulder arthroplasty (TSA) is the surgical treatment of choice for patients suffering from glenohumeral OA (4, 5). The aim of TSA is to relieve pain and thereafter improve physical function (6-9). Although the incidence of TSA is rising, and 70% of patients report that they are very satisfied with their postoperative results (10), the proportion of patients living with an unsatisfactory shoulder arthroplasty is largely unknown (11).

In hip and knee OA exercise is recommended as the first-line treatment (4). The effectiveness of exercise and the effectiveness of TSA in patients with glenohumeral OA is unknown, as no randomized trials have directly compared TSA to a non-surgical treatment (5). In order to provide a trustworthy and evidence-based foundation for clinical decisions it is important to conduct a randomized controlled trial where surgical treatment is compared to non-surgical treatment in patients with glenohumeral OA.

Date: 02.07.2024

Version: 1.0

The primary aim of this trial is to examine if surgical treatment followed by standard care is

superior to a 12-week exercise programme in patients with primary glenohumeral OA. The

primary outcome is the Western Ontario Osteoarthritis of the Shoulder index score (WOOS),

measured 12 months after initiating the treatment. The primary hypothesis is that surgical

intervention is superior to the exercise intervention at 12 months (1).

The key secondary objectives are (1):

1. To investigate the effectiveness of total anatomical shoulder arthroplasty followed by

standard rehabilitation compared to a 12-week physiotherapist-supervised exercise

programme, on (1) pain intensity, (2) activities of daily living, (3) use of analgesics and

(4) shoulder-related quality of life in patients with glenohumeral OA.

2. To investigate the safety of total anatomical shoulder arthroplasty followed by standard

rehabilitation compared to a 12-week physiotherapist-supervised exercise programme

on occurrence of adverse events from baseline to 12 months after initiating the

treatment, in patients with glenohumeral OA.

Exploratory objectives:

1. To investigate the external validity of the randomised controlled trial on total

anatomical shoulder arthroplasty and physiotherapist-supervised exercise in patients

glenohumeral OA by comparing patient characteristics and patient-reported WOOS

scores from baseline to 12 months after initiating the treatment, in patients included in

the randomised controlled trial versus those declining to participate but included in the

follow-up cohort.

2. To investigate objectively measured physical upper extremity activity level from

baseline to 12 months using tri-axial (Axivity, UK) accelerometers, in patients with

glenohumeral OA eligible for total anatomical shoulder arthroplasty.

3. To assess the cost-utility of total anatomical shoulder arthroplasty followed by standard

care compared to a 12-week physiotherapist-supervised progressive exercise

programme on quality-adjusted life years (QALYs) gained from baseline to 12 months

after initiating the treatment, in patients with glenohumeral OA.

**SECTION 3: STUDY METHODS** 

**Trial Design** 


The PROACT trial is a multicenter randomized controlled and investigator blinded trial, the reporting of the trial will follow the "Consolidated Standards of Reporting Trials" (CONSORT) statement (12). Patients are recruited from the orthopaedic departments at Aarhus University Hospital, Aalborg University Hospital, Viborg Regional Hospital and Silkeborg Regional Hospital in Denmark, at Tampere University Hospital, Central Finland Hospital in Finland and Oslo University Hospital in Norway.

The Statistical Analysis Plan (SAP) is reported in accordance with the "Guidelines for the Content of Statistical Analysis Plan in Clinical Trials" (13).

The PROACT trial is registered at <a href="www.clincaltrials.gov">www.clincaltrials.gov</a> with the number NCT04845074. The Central Denmark Region Committee on Biomedical Research Ethics (Journal No 1-10-72-29-21) and the Danish Data Protection Agency (Journal No 1-16-02-199-21), The Regional Ethics Committee of the Expert Responsibility area of Tampere University Hospital (ref ETL R21089) and The Regional Committee for Medical and Health Research Ethics Region South-East Norway (Ref. 269784) have approved the trial.

#### Randomisation

The included patients will be randomised with a 1:1 allocation to TSA or exercise after their baseline assessment. The randomisation is stratified by recruitment site with randomly selected block sizes and done by a computer-generated list of random numbers using the randomization tool in Research Electronic Data Capture (REDCap), developed by an independent data manager (14). During the trial period administrators of the randomisation procedure are blinded to block sizes and randomisation sequence at all times.

## Sample Size

The sample size is based on the expected between group difference in the WOOS end scores. The WOOS score 1 year after TSA surgery was 84.6 points in the Danish Shoulder Arthroplasty Registry in 2020 (7). The WOOS score after completing this exercise intervention in a feasibility study was 67 points (15). The assumed common SD was 27.1. The required power was set to 80%. Given a power of 0.80 to detect a difference between the two groups and using a two-sided significance level  $\alpha$ =0.05, the estimated sample of each intervention group is 39 patients. Allowing for possible crossovers, loss-to follow-up and drop-outs the total number of patients in each group is 51 (1).

## Framework

The overall objective of the trial is to determine whether surgical intervention results in a clinically and statistically significant greater improvement compared to exercise on WOOS, Disabilities of the Arm, Shoulder and Hand (DASH) (16), patient-reported pain intensity at rest, during activity, and nightly pain using the 100 mm VAS, the use of analgesics during the last week (paracetamol, NSAID, opioids) and adverse events. The primary hypothesis is that surgical intervention is superior to the exercise intervention at 12 months.

## Blinded interpretation of the results

The blinded interpretation will be of the intention-to-treat analysis. The blinded analysis involves the primary outcome and key secondary outcomes. The principal investigator (JBL) will export data from REDCap and deliver the blinded dataset for analysis to the statistical analysist (AR). The senior statistician (EP) will supervise the analysis. The blinded results from the analysis of treatment A compared with treatment B will be presented to the project group followed by the development of the blinded interpretation. Interpretation version 1 assumes that group A had surgery, while interpretation 2 assumes that group A performed exercise. A draft of the blinded interpretation will be sent for approval by all co-authors. No other outcomes will be analyzed prior to an agreement of the blinded interpretation by all co-authors. All other analyses described in this document will be performed after the blinded interpretation is published (17).

# Statistical interim analysis and stopping guidance

There has not been planned any formal statistical interim analysis for the PROACT trial. The final deadline for patient recruitment was a priori set to April 2024 but has since been moved to November 2024 due to delays in recruitment.

## Timing of final analysis

The final analysis for the primary outcome, the end scores on WOOS at 12 months, will be performed after the last follow-up assessment at 12-months. The main publication of the trial will be prepared when these data are available.

In addition, papers on 2-, 5-, and 10-years follow-up will be performed, when these follow-up

assessments are available.

Timing of outcome assessments

The trial consists of six time points; baseline, 12-weeks, 12-months, 2 years, 5 years and 10

years. An overview of the assessments and procedures has been presented in the protocol

(Table 1).

**SECTION 4: STATISTICAL PRINCIPLES** 

Confidence intervals and P values

For the primary outcome the statistical tests will be two-sided and a p-value <0.05 will be

considered statistically significant. Confidence intervals will be 95% (95% CI) and two-

sided. For the secondary outcomes the use of p values will be interpreted with care (18).

Adherence and protocol deviations

Adherence is defined as the ability to follow the allocated treatment. For the exercise group

adherence is related to the number of attended supervised exercise sessions, good adherence

has been predefined as participation in at least 70% of the supervised exercise sessions,

during the first 12-weeks. Table 7 illustrates this.

There are predefined protocol deviations regarding adherence:

1. Patients randomized to exercise undergoing TSA in the follow-up period

2. Patients randomized to TSA not undergoing TSA in the follow-up period

**Analysis populations** 

The primary analysis will be based on the Intention to Treat (ITT) principle. Patients allocated

to a treatment group (TSA or exercise) should be followed up, assessed and analysed as

members of that group, regardless of their adherence to the planned course of treatment.

Response to treatment will be described for both treatment groups, regardless of their

adherence to the planned course of treatment.


Version: 1.0

A per protocol analysis will be conducted with patients in the surgical group undergoing

surgery and for the exercise groups patients with a good adherence to the exercises are included.

Poor adherence is defined as participating in less than 70% of the supervised exercise sessions.

Another per protocol analysis will be of patients undergoing surgery regardless of

randomization.

Lastly four as-treated analysis will be performed in which patients will be analyzed based on

their adherence to the randomized treatment expecting four groups: (1) patients randomized

to TSA and getting TSA, (2) patients randomized to exercise without undergoing TSA in the

follow-up period, (3) patients randomized to exercise undergoing TSA in the follow-up

period, (4) patients randomized to TSA not undergoing TSA in the follow-up period. One as

treated analysis will be done on TSA patients versus good exercise adherence versus poor

exercise adherence. And one as treated analysis on TSA patients randomized to TSA versus

crossover TSA patients versus good exercise adherence versus poor exercise adherence.

**SECTION 5: TRIAL POPULATION** 

Screening data

At all hospitals patients eligible for TSA will be screened for the inclusion and exclusion

criteria. If they fulfil the criteria, they will be invited to participate. The number of patients

who do not meet the criteria and the reason for ineligibility will be reported in a CONSORT

flow chart (Figure 1).

**Eligibility** 

Patients fulfilling the in- and exclusion criteria and are willing to participate are eligible for

the PROACT trial. The inclusion criteria are:

Inclusion criteria:

1. Patients  $\geq$ 55 years

2. Moderate to severe primary OA of the glenohumeral joint (Osteophyte larger than 3

mm, according to Samilson and Prieto (Samilson et al. 1983)

3. Eligible for surgery with standard TSA


#### Exclusion criteria:

- 1. Surgical need for bone graft or use of augmented glenoid component
- 2. Previous shoulder fracture (fracture of the proximal humerus or glenoid fracture)
- 3. Planned other upper extremity surgery within six months
- 4. Rheumatoid arthritis or other types of arthritis not diagnosed as primary glenohumeral OA
- 5. Cancer diagnosis and actively receiving chemo-, immuno-, or radiotherapy
- 6. Neurological diseases affecting shoulder mobility (e.g., disability after previous stroke, multiple sclerosis, Parkinson's, Alzheimer's disease)
- 7. Other reasons for exclusion include mentally unable to participate or planned absence for more than 14 days in the first 3 months after baseline test
- 8. Unable to communicate in the respective languages of the participating countries.

#### Recruitment

The CONSORT flowchart will present the number of patients screened, excluded (with reasons), eligible for inclusion, randomized, receiving allocated treatment, withdrawals (with reasons), lost to follow-up (with reasons), included in the ITT analysis, included in the per protocol analysis.

#### Withdrawal/follow-up

Throughout the trial period the patients are allowed to withdraw from the study at any time. Patients who decide to withdraw will be encouraged to continue in the study as if they have received the intervention. Withdrawal will be classified into two options; (1) complete withdrawal from the study with no further follow-up and data-collection, (2) consent to follow-up assessments and data-collection. The number of withdrawals and the timing of withdrawal will be presented in the CONSORT flowchart (with reasons).

# **Baseline patient characteristics**

Baseline characteristics will be presented as seen in Table 2. Categorical variables will be presented as numbers and percentages. Continuous variables will be presented as mean with

Version: 1.0

standard deviation (SD), if normally distributed and ad median with interquartile range (IQR) if not normally distributed. No tests of significance will be conducted for the baseline characteristics, imbalances of importance will be noted. Baseline and follow-up values for the primary and secondary outcomes will be presented as part of the analysis, as seen in Table 3.

**SECTION 6: ANALYSIS** 

**Outcome definitions** 

The Western Ontario Osteoarthritis of the Shoulder index score (WOOS)

The primary outcome will be presented as the between group difference on the 12-month follow-up score. WOOS is a valid and reliable patient-reported questionnaire assessing shoulder pain and function in a total raw score ranging from 0-1900, raw scores can be converted to a score from 0-100, where 0 indicates severe problems and 100 indicates no problems.

**Key secondary outcomes** 

Disabilities of the Arm, Shoulder and Hand (DASH) (Lindenhovius et al. 2008); patient-reported pain intensity at rest, during activity, and nightly pain using the 100 mm VAS; the use of analgesics during the last week (paracetamol, NSAID, opioids); serious adverse events and adverse events.

**Analysis methods** 

Descriptive statistics will be presented as means with standard deviation (SD) for all normally distributed continuous variables. Continuous variables that do not follow a normal distribution will be presented as median with interquartile ranges. Normal distribution will be determined by visual inspection of QQ-plots and histograms. Categorical outcomes will be presented as numbers with percentages.

The primary comparison in WOOS between groups will be conducted using a linear mixed model. Intervention group and time (3 months, 12 months) will be included as fixed effects and patient as random. Baseline score, sex, age and study site will also be included as fixed covariates. Interaction between study group and time will be included in the model to estimate treatment effect at each time point. 95% confidence intervals are estimated for each time point.

Date: 02.07.2024

Version: 1.0

Due to the repeated mixed model analysis no missing data imputation will be conducted. A

sensitivity analysis will be done using an analysis of covariance (ANCOVA) including baseline

score, sex, age and study site as covariates with the same ITT approach for time (3 months and

12 months) separately.

Analysis for patient-reported DASH, pain intensity at 3 and 12 months will be analysed similar

to the primary comparison. For binary variables (ie. the use of analgesics and adverse events)

we use proportions to describe the number of events. For each binary outcome an unadjusted

risk difference in proportions with 95% confidence interval of outcomes between study groups.

Table 3 illustrates the primary analysis.

Response to treatment for the WOOS change score from baseline to 12 months and 3 months

follow-up will be computed for each patient in both treatment groups. Response to treatment

will be presented dichotomized (i.e. responder and non-responder) as number and percentage.

The patients will be classified as a responder if they reach a minimal important change of 13.3

points or more from baseline to 12 months follow-up (19).

Missing data

As stated above, imputations will not be applied in this study due to the repeated mixed model

analysis. Each randomized patient will be included in the intention-to-treat analysis with the

collected data. In an attempt to collect data from all randomized patients, patients deciding to

withdraw from the study, are still encouraged to attend the follow-up test.

Harms

Adverse and serious adverse events will be presented as number and percentage for each

event.

Statistical software

All statistical analysis will be conducted using the statistical software program R (R

Foundation for Statistical Computing, Vienna, Austria) (20).


#### REFERENCES

1. Beck Larsen J, Thillemann TM, Launonen AP, Østergaard HK, Falstie-Jensen T, Reito A, et al. Study protocol: Prosthesis versus Active (ProAct) exercise program in patients with glenohumeral osteoarthritis — a multicenter, randomized controlled trial. Acta Orthop. 2022;93:303-16.

- 2. Ansok CB, Muh SJ. Optimal management of glenohumeral osteoarthritis. Orthop Res Rev. 2018;10:9-18.
- 3. Macias-Hernandez SI, Morones-Alba JD, Miranda-Duarte A, Coronado-Zarco R, Soria-Bastida MLA, Nava-Bringas T, et al. Glenohumeral osteoarthritis: overview, therapy, and rehabilitation. Disabil Rehabil. 2017;39(16):1674-82.
- 4. Roos EM, Juhl CB. Osteoarthritis 2012 year in review: rehabilitation and outcomes. Osteoarthritis Cartilage. 2012;20(12):1477-83.
- 5. Craig RS, Goodier H, Singh JA, Hopewell S, Rees JL. Shoulder replacement surgery for osteoarthritis and rotator cuff tear arthropathy. Cochrane Database Syst Rev. 2020;4:Cd012879.
- 6. Rasmussen JV, Olsen BS. The Danish Shoulder Arthroplasty Registry. Obere Extrem. 2019;14(3):173-8.
- 7. Registry) YrDSA, Register) OÅDS. Yearly report (Danish Shoulder Arthroplasty Registry)
- Original: Årsrapport (Dansk Skulderalloplastik Register). 2020;2021(24th of February).
- 8. Rasmussen JV, Polk A, Brorson S, Sørensen AK, Olsen BS. Patient-reported outcome and risk of revision after shoulder replacement for osteoarthritis. 1,209 cases from the Danish Shoulder Arthroplasty Registry, 2006-2010. Acta Orthop. 2014;85(2):117-22.
- 9. Rasmussen JV, Amundsen A, Sorensen AKB, Klausen TW, Jakobsen J, Jensen SL, et al. Increased use of total shoulder arthroplasty for osteoarthritis and improved patient-reported outcome in Denmark, 2006-2015: a nationwide cohort study from the Danish Shoulder Arthroplasty Registry. Acta Orthop. 2019;90(5):489-94.
- 10. Sowa B, Thierjung H, Bülhoff M, Loew M, Zeifang F, Bruckner T, et al. Functional results of hemi- and total shoulder arthroplasty according to diagnosis and patient age at surgery. Acta Orthop. 2017;88(3):310-4.
- 11. Craig RS, Lane JCE, Carr AJ, Furniss D, Collins GS, Rees JL. Serious adverse events and lifetime risk of reoperation after elective shoulder replacement: population based cohort study using hospital episode statistics for England. BMJ. 2019;364:1298.
- 12. Moher D, Hopewell S, Schulz KF, Montori V, Gøtzsche PC, Devereaux PJ, et al. CONSORT 2010 Explanation and Elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010;340:c869.
- 13. Gamble C, Krishan A, Stocken D, Lewis S, Juszczak E, Doré C, et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. JAMA. 2017;318(23):2337-43.
- 14. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009;42(2):377-81.
- 15. Beck Larsen J, Østergaard HK, Thillemann TM, Falstie-Jensen T, Urup Tønning L, Noe S, et al. Are progressive shoulder exercises feasible in patients with glenohumeral osteoarthritis or rotator cuff tear arthropathy? Pilot and Feasibility Studies. 2022.

- 16. Lindenhovius A, Buijze G, Kloen P, Ring D. Correspondence Between Perceived Disability and Objective Physical Impairment After Elbow Trauma. J Bone Joint Surg Am. 2008;90:2090-7.
- 17. Järvinen TL, Sihvonen R, Bhandari M, Sprague S, Malmivaara A, Paavola M, et al. Blinded interpretation of study results can feasibly and effectively diminish interpretation bias. J Clin Epidemiol. 2014;67(7):769-72.
- 18. Harrington D, D'Agostino RB, Sr., Gatsonis C, Hogan JW, Hunter DJ, Normand ST, et al. New Guidelines for Statistical Reporting in the Journal. N Engl J Med. 2019;381(3):285-6.
- 19. Larsen JB, Thillemann TM, Launonen AP, Østergaard HK, Falstie-Jensen T, Sumrein B, et al. Minimal important change of the Western Ontario Osteoarthritis of the Shoulder (WOOS) index in patients with glenohumeral osteoarthritis and rotator cuff tear arthropathy. Archives of Orthopaedic and Trauma Surgery (in review). 2024.
- 20. R Core Team. R: A language and environment for statistical computing.: R Foundation for Statistical Computing, Vienna, Austria.; 2021 [Available from: https://www.R-project.org/.

Figure 1 Expected enrolment, randomization, intervention, and follow-up. Total shoulder arthroplasty (TSA).



Table 1. Assessments and procedures.

| | Baseline | Surgery | 3 m | 12 m | 2 y | 5 y | 10 y |
|---|---|---|---|---|---|---|---|
| Baseline characteristics | | | | | | - | |
| Sex | X | | | | | | |
| Age | X | | | | | | |
| Height | X | | | | | | |
| Weight | X | | | | | | |
| Hand dominance | X | | | | | | |
| Duration of shoulder symptoms | X | | | | | | |
| Marital status | X | | | | | | |
| Educational level | X | | | | | | |
| Employment status | X | | | | | | |
| Alcohol intake | X | | | | | | |
| Smoking behaviors | X | | | | | | |
| Comorbidities | X | | | | | | |
| Surgery information | | | | | | | |
| X-ray and surgeon appointment | X | | | | | | |
| Surgery report (only surgical group) | | X | $X^*$ | $X^*$ | | | |
| CT | X | | | | | | |
| Patient reported outcomes | | | | | | | |
| WOOSa | X | | X | X | X | X | X |
| DASH <sup>b</sup> | X | | X | X | X | X | X |
| EQ-5D-5L° | X | | X | X | X | X | X |
| iPCQ d | | | X | X | | | |
| VASe | X | | X | X | X | X | X |
| Physical activity | | | | | | | |
| Tri-axial accelerometry | X | | | X | | | |
| Treatment related variables | | | | | | | |
| Adverse events <sup>f</sup> | | | X | X | X | X | X |
| Serious adverse events <sup>f</sup> | | | X | X | | | |
| Training-compliance | | | X | | | | |
| Pain before exercise and at the end of | | | 37 | | | | |
| exercise for the exercise group using NRSg | | | X | | | | |
| Other shoulder related treatments | X | | X | X | | | |
| Analgesic consumption in last week | X | | X | X | X | X | X |
| Crossover | | | X | X | X | X | X |

m = months. y = years. \*X-ray at 3 months for the surgical group only to assess adverse events. a the Western Ontario Osteoarthritis of the Shoulder index (WOOS). Disabilities of the Arm, Shoulder and Hand (DASH). European Quality of life 5 Dimensions with 5 Levels (EC-5D-5L). Productivity Costs Questionnaire (iPQC) only in Denmark. Visual Analogue Scale will be at rest, during activity and at night. Described in "Adverse events". Numeric Rating Scale will be used at the supervised exercise sessions to determine pain at rest before and after the session.

Table 2: Baseline characteristics for the two intervention groups

| | TSA group | Exercise group |
|---|---|---|
| | n= | n = |
| Gender, n (%) female | | |
| Age, mean (SD) years | | |
| Body mass index, mean (SD) kg/m <sup>2</sup> | | |
| Handedness, n (%) right | | |
| Affected shoulder, n (%) right | | |
| Duration of shoulder symptoms, n (%) | | |
| 6-12 months | | |
| 1-2 years | | |
| 2-5 years | | |
| More than 5 years | | |
| Previous treatment in the affected shoulder, n (%) yes | | |
| Exercise and/or physiotherapy | | |
| Pharmacological treatment | | |
| Surgical treatment | | |
| Civil status, n (%) | | |
| Living alone | | |
| Living with someone | | |
| Not informed | | |
| Educational level, n (%) | | |
| Low | | |
| Medium | | |
| High | | |
| Employment status, n (%) | | |
| Employed | | |
| Outside the labor market | | |
| In activation, sick leave, available, etc. | | |
| Retired | | |
| Alcohol consumption, n (%) | | |
| Under 2 items per week | | |
| 2-7 items per week | | |
| 8-14 items per week | | |
| 15-21 items per week | | |
| Over 21 items per week | | |
| Smoking behaviour, n (%) | | |
| Never smoked | | |
| Quit smoking | | |
| Sometimes | | |
| Daily | | |
| Co-morbidities, n (%) yes | | |

Table 3: Intention to treat analysis and per protocol analysis of the between group difference for the surgical group and exercise group in end-scores one year after intervention.

| | | - | Intention | -to-treat an | alysis | | |
|---|---|---|---|---|---|---|---|
| | TSA | | | | Exercise | Improvement<br>between the two<br>groups | |
| | Baseline | Three | One | Baseline | Three | One | Adjusted |
| | | months | year | | months | year | |
| WOOS | | | | | | | |
| DASH | | | | | | | |
| Pain at rest | | | | | | | |
| Pain during | | | | | | | |
| activity | | | | | | | |
| Pain at night | | | | | | | |
| Use of | | | | | | | |
| analgesics* | | | | | | | |
| Adverse events* | | | | | | | |
| | | | Per-pr | otocol analy | ysis | L | |
| | | TSA | | | Exercise | | Improvement |
| | | | | | | | between the two |
| | | | | | | | groups |
| | Baseline | Three | One | Baseline | Three | One | Adjusted |
| | | months | year | | months | year | |
| WOOS | | | | | | | |
| DASH | | | | | | | |
| Pain at rest | | | | | | | |
| Pain during | | | | | | | |
| activity | | | | | | | |
| Pain at night | | | | | | | |
| Use of | | | | | | | |
| analgesics* | | | | | | | |
| Adverse events* | | | | | | | |

Higher scores indicate desired (better) treatment outcome for WOOS. For the other outcomes lower scores indicate desired (better) treatment outcome.

<sup>\*</sup>Analysed with risk difference, use of analgesics (yes/no), adverse events (yes/no).

Table 4: As treated analysis of the between group difference for the surgical group and

exercise group in end-scores one year after intervention.

| exercise group | TS | | | | ercise | | | oss-ov | | No | No<br>treatment | | Improvements between the four groups |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | В | 3M | 1 <b>Y</b> | В | 3M | 1Y | В | 3M | 1Y | В | 3M | 1 <b>Y</b> | Adjusted |
| woos | | | | l | | | <u> </u> | | | | | | L |
| DASH | | | | | | | | | | | | | |
| Pain at rest | | | | | | | | | | | | | |
| Pain during activity | | | | | | | | | | | | | |
| Pain at night | | | | | | | | | | | | | |
| Use of analgesics* | | | | | | | | | | | | | |
| Adverse events* | | | .1. 43 | | | | | | | | | | |

B=Baseline, 3M=Three months, 1Y=One year

Table 5: Usage of painkillers

| | TSA group | | | Exercise group | | |
|---|---|---|---|---|---|---|
| | Baseline | Three months | One year | Baseline | Three | One year |
| | | | | | months | - |
| Use of painkillers, n (%) yes | | | | | | |
| Type of painkillers, n (%) | | | | | | |
| Paracetamol | | | | | | |
| NSAID | | | | | | |
| Morfin/opiods | | | | | | |
| Other painkillers | | | | | | |
| Usage of painkillers, n (%) | | | | | | |
| Never | | | | | | |
| Monthly | | | | | | |
| Weekly | | | | | | |
| Daily | | | | | | |

**Table 6: Adverse and serious adverse events** 

| | TSA group | Exercise group |
|-----------------------------------------------|-----------|----------------|
| Adverse events, n (%) | | |
| Postoperative infections | | |
| Instability | | |
| Periprosthetic fracture | | |
| Loosening | | |
| Humeral component | | |
| Glenoid component | | |
| Both | | |
| Injuries related to the exercise intervention | | |
| Serious adverse events, n (%) | | |
| Death | | |
| Embolism | | |
| Liver failure | | |
| Renal failure | | |

<sup>\*</sup>Serious adverse events resulting in the need for hospitalization or death in the first 4 weeks after surgery. Adverse events that occurred between baseline and 12 months follow-up but did not necessarily have a causal relationship between the treatments.

Table 7: Adherence to randomized treatment

follow-up period, n (%)

Exercise group Training adherence Showed up for supervised sessions within the first three months of exercise, mean Participated in at least 70% of supervised sessions within the first three months of exercise, n (%) Number of self-reported exercise sessions within the first three months of exercise, mean (SD) Completed three or more exercise sessions per week within the first three months of exercise, n (%) Completed 4 booster sessions, n (%) Number of self-reported exercise sessions from three months to one year, mean (SD) Completed three or more exercise sessions per week from three months to one year, n (%) Number of patients randomized to exercise undergoing surgery in the follow-up period, n (%) Surgical group Surgical adherence Number of patients randomized to surgery electing not to undergo surgery in the